CLINICAL TRIAL: NCT04119830
Title: A Phase IIa Study of Rintatolimod Plus Pembrolizumab in Refractory Metastatic Colorectal Cancer
Brief Title: Rintatolimod and Pembrolizumab for the Treatment of Refractory Metastatic or Unresectable Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: implementation issues
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 74118; NCI-2019-06440 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 74118 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-10-07; First posted 2019-10-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Metastatic Colorectal Adenocarcinoma; Microsatellite Stable; Mismatch Repair Proficient; Refractory Colorectal Adenocarcinoma; Stage III Colorectal Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8; Unresectable Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pembrolizumab; poly(I).poly(c12,U)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (rintatolimod, pembrolizumab) (Experimental): Patients receive rintatolimod IV over 30 minutes on days 1-3 and pembrolizumab IV over 30 minutes on day 3. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Beginning in cycle 4, patients receive rintatolimod IV over 30 minutes and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 24 months from the first dose in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Other: Questionnaire Administration; Drug: Rintatolimod

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Questionnaire Administration — Ancillary studies
Drug: Rintatolimod — Given IV
  Other Names: Ampligen; Atvogen

SUMMARY:
This phase IIa trial studies how well rintatolimod and pembrolizumab works in treating patients with colorectal cancer that does not respond to treatment (refractory), has spread to other places in the body (metastatic), or otherwise cannot be removed by surgery (unresectable). Rintatolimod is an immuno-oncology agent that can stimulate the immune system. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving rintatolimod and pembrolizumab together may work better than standard of care in treating patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the objective response rate of patients with metastatic colorectal cancer (mCRC) treated with rintatolimod + pembrolizumab.

SECONDARY OBJECTIVES:

I. Establish the adverse event profile of combining rintatolimod and pembrolizumab.

II. Estimate the median progression free survival and overall survival of patients with mCRC treated with rintatolimod and pembrolizumab.

III. Determine the immune objective response rate of patients with mCRC treated with rintatolimod + pembrolizumab.

EXPLORATORY OBJECTIVES:

I. Assess modulation of the levels of CD8alpha expression and cytotoxic T-lymphocyte (CTL) density pre- and post-therapy.

II. Assess chemokine levels in the tumor microenvironment and peripheral blood, including effector T cell (Teff)-attracting and regulatory T cell (Treg)-favoring chemokines.

III. Characterize the fecal microbiotic profile and correlate those results with antitumor immune responses.

OUTLINE:

Patients receive rintatolimod intravenously (IV) over 30 minutes on days 1-3 and pembrolizumab IV over 30 minutes on day 3. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Beginning in cycle 4, patients receive rintatolimod IV over 30 minutes and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 24 months from the first dose in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days, and every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven colorectal adenocarcinoma which is metastatic or otherwise unresectable
* Microsatellite stable/mismatch-repair proficient (by immunohistochemistry [IHC] and/or polymerase chain reaction [PCR])
* Progression following: a fluoropyrimidine, oxaliplatin, irinotecan, and anti-EGFR targeted therapy (if anti-EGFR therapy is appropriate), bevacizumab (if appropriate)

  * NOTE: Patients who could not tolerate standard agents because of unacceptable, but reversible, toxicity necessitating their discontinuation will be allowed to participate
* Amenable to undergoing serial tumor biopsy (x 2). NOTE: patients with inaccessible lesions, where the investigator deems biopsy to be unsafe or where biopsy is otherwise contraindicated, are still eligible to enroll, with review and approval of the principal investigator (PI)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil (ANC) count >= 1500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9 g/dL
* Serum or plasma creatinine =< 1.5 X upper limit of normal (ULN) or measured or calculated creatinine clearance by Cockcroft Gault Equation >= 30 ml/min for subjects with creatinine levels > 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN or (=< 5 x ULN if the patient has liver metastases)
* Bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN
* International normalized ratio (INR) or prothrombin time (PT): =< 1.5 unless participant is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT): =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria present
* Female participants of childbearing potential are to have a negative serum pregnancy test
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment
* A male participant must agree to use an adequate method of contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to start of study treatment
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette?Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of systemic immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has a known additional malignancy that is progressing or in the opinion of the investigator is likely to interfere with properly assessing treatment efficacy. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Have a severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Has previously received rintatolimod, poly-ICLC or derivatives
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Woman of childbearing potential who has a positive urine pregnancy test within 72 hours prior to start of study treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV), unless on highly active antiretroviral therapy (HAART) with undetectable viral load
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected) infection
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator?s opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | At 6 months following completion of enrollment (at 24 months)
  Determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and estimated using a 90% confidence interval obtained using Jeffrey?s prior method.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Toxicities and adverse events (according to Common Terminology Criteria in Adverse Events [CTCAE] version 5.0) will be summarized by attribution and grade using frequencies and relative frequencies.
Median progression free survival | From the time of first dosing of study treatment combination to documented disease progression by RECIST 1.1, assessed up to 2 years
  Will be summarized using standard Kaplan-Meier methods; where estimates of median survival and 6/12-month survival rates will be obtained with 95% confidence intervals.
Overall survival | From the time of first dosing of study treatment combination to time of death or initiation of a new therapy, whichever occurs first, assessed up to 2 years
  Will be summarized using standard Kaplan-Meier methods; where estimates of median survival and 6/12-month survival rates will be obtained with 95% confidence intervals.
Objective response rate | Up to 2 years
  Determined by immune-modified (i)RECIST and estimated using a 90% confidence interval obtained using Jeffrey?s prior method.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Fountzilas, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States